CLINICAL TRIAL: NCT04369118
Title: Efficacy Study of a Selective Chest Wall Restriction Belt in Postoperative of Lung Resection. A Multicenter, Prospective, Controlled, Randomized Study With Stratification on the Surgical Approach, Open With a Blind Analysis
Brief Title: Efficacy Study of a Selective Chest Wall Restriction Belt in Postoperative of Lung Resection
Acronym: CTS-POP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Clinical Investigation Centre for Innovative Technology Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 38RC19.102
Record Dates: First submitted 2020-03-10; First posted 2020-04-30 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Lung Cancer
Keywords: chest wall restriction; usability; lung surgery; medical device; pain; cough; expectoration
MeSH Terms: conditions — Lung Neoplasms; Pain; Cough

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional follow-up+chest wall restriction belt (Experimental): Patients in this group benefit from conventional post-operative follow-up and wear the selective chest wall restriction belt in parallel. Patients in this group benefit from conventional post-operative follow-up . From Day 1 to Month 1
  Interventions: Procedure: Conventional follow-up; Device: Conventional follow-up+chest wall restriction belt
- conventional postoperative follow-up (Active Comparator): Patients in this group benefit from conventional post-operative follow-up . From Day 1 to Month 1
  Interventions: Procedure: Conventional follow-up

INTERVENTIONS:
Procedure: Conventional follow-up — Patients in this group benefit from conventional post-operative follow-up
Device: Conventional follow-up+chest wall restriction belt — Patients in this group benefit from conventional post-operative follow-up. The patient wear the selective chest wall restriction belt from Day 2 (after surgery) until he ceases to need it.
  Arms: Conventional follow-up+chest wall restriction belt

SUMMARY:
The objective of this study is to evaluate the efficacy of a new medical device in post-surgery of lung resection. The principle of this new device is based on selective chest wall restriction. This new modality of chest wall restriction is evaluated on patients in post-surgery for lung cancer.

The hypothesis is that the use of this medical device would reduce the postoperative pain and increase the efficacy of cough and expectoration. The evolution of the operated patient would be better.

DETAILED DESCRIPTION:
The present study is the first evaluation of the efficacy of a selective chest wall restriction belt.

The efficacy will be estimate on forced expiratory volume in one second (FEV1) at D3 by comparing 2 groups: a control group of patients with conventional follow-up and an experimental group of patients with conventional follow-up and a daily wear of the selective chest wall restriction belt after surgery.

ELIGIBILITY:
Inclusion Criteria :

* Patients with segmentectomy or lobectomy for lung cancer or lung cancer suspicious,
* Surgical approach : video-assisted thoracic surgery (VATS) or thoracotomy,
* Patients affiliated to social security or similarly regime,
* Patients who gave their consent to participate in the study.

Exclusion Criteria :

* Patients with outcomes of the pulmonary function test at the preoperative assessment : forced expiratory volume in one second (FEV1) or diffusing capacity of the lung for carbon monoxide (DLCO) > 45% predicted post-operative values and VO2max (maximal oxygen consumption) between 10 and 12 ml/kg/min,
* Patients with a waist size > 120 cm
* Patients with medical treatment for chronic pain (neuropathic pain,…)
* Patients with tuberculosis or other pulmonary infectious pathology proven (aspergillosis, lung abscess, actinomycosis,…),
* Patients carrying a resistant germs or extended-spectrum beta-lactamase (ESBL),
* Paraplegic patients
* Patients with a diagnosed, progressive and/or uncontrolled neurological disease
* Patients with a progressive psychosis or a serious psychotic history (hospitalization)
* Patients who are in exclusion period of another interventional study
* Protected person referred to in Articles L1121-5 to L1121-8 of the Code of Public Health

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Comparison of forced expiratory volume in one second (FEV1) between the two groups. | 3 days
  Comparisons of forced expiratory volume in one second (FEV1) between the two groups at Day 3. The value of FEV1 is standardized with pre-operative one.

SECONDARY OUTCOMES:
Comparisons of pulmonary function test between the two groups | 1 month
  Comparisons of pulmonary function test ( forced expiratory volume in one second (FEV1), Forced vital capacity (FVC)) between the two groups. They are expressed as Liters. Before surgery, all days from Day 2 to the patient's exit from hospital (max Day 6) and at the follow-up visit at Month 1. Each value is standardized with pre-operative one.
Comparisons of Peak expiratory flow at cough between the two groups | 1 month
  Comparisons of Peak expiratory flow at cough (PEF) between the two groups. It is expressed as Liters per second. Before surgery, all days from Day 2 to Day 6 and at the follow-up visit at Month 1. Each value is standardized with pre-operative one.
Pain evaluation at rest and during cough: ENS scale | 1 month
  The patient pain is evaluated using the ENS (Echelle Numérique Standard; standard digital scale, score between 0 to 10) for the two groups. The pain is evaluated all days from Day 2 to the patient's exit from hospital, at the weekly phone follow-up until Month 1 and at the follow-up visit at Month 1.
Qualification of cough | 10 days
  The cough is classified with this scale : 0-dry cough; 1-productive cough without expectoration; 2-productive cough with expectoration; 3-productive cough with important and/or difficult expectoration. It's qualified for the two groups all days from Day 2 to the patient's exit from hospital.
Characterization of analgesic treatment. | 1 month
  The analgesic drugs are characterized by their class, dose and number of dose taken in the two groups. These elements are evaluated all days from Day 2 to the patient's exit from hospital, at the weekly phone follow-up until Month 1 and at the follow-up visit at Month 1.
Identification of using aerosol therapy, antibiotic therapy and loco-regional anaesthesia | 1 month
  Use of aerosol therapy (yes/no) and class of drugs. Use of antibiotic therapy (yes/no), type of drugs and expected duration of treatment. Use of loco-regional anaesthesia (yes/no), modality of administration and type of drugs. These elements are evaluated all days from Day 2 to the patient's exit from hospital, at the weekly phone follow-up until Month 1 and at the follow-up visit at Month 1.
Number and classification of post-surgery complications | 1 month
  Number and classification of post-surgery complications.For the two groups from Day 1 to the follow-up visit at Month 1.
The length of hospital stay | 10 days
  The length of hospital stay in days for the two groups.
Quantification of the quality of life evaluated with the EQ-5D-5L questionnaire | 1 month
  The EQ-5D is a generic preference-based measure that indirectly measures the utility for health that generates an index-based summary score based upon societal preference weights. The EQ-5D-5L consists of 6 items that cover 5 main domains (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) and a general visual analog scale (VAS) for health status. Each item has 5 response levels ranging from level 1 (no problem or none) to level 5 (unable to perform activity). The VAS ranges from 0 (worst health status) and 100 (best health status). Comparison between the two groups preoperatively, at the patient's exit from hospital, at Day 15 during the phone follow-up and at the follow-up visit at Month 1.
Consumption of hospital care | 1 month
  Comparions of the number of the consumption of hospital care (medical acts and consultations, rehospitalization) between the two groups from Day 1 to the follow-up visit at Month 1.
Evaluation of medical device usability for patient | 1 month
  Only for the medical device's group.
  1. Qualitative questionnaire specifically created about efficacy and acceptability of the medical device at the patient 's exit from hospital. This questionnaire uses Likert scale from 0 to 10 to evaluate each use step of the medical device, closed-ended questions and open questions for comments. A descriptive analysis will done with the answers
  2. Closed-ended questions will be asked in a questionnaire specifically created about acceptability and use of the medical device. A descriptive analysis will done with the answers and will be asked during the weekly phone follow-up.
Evaluation of medical device usability for caregivers | 1 month
  Only for the medical device's group. This questionnaire uses Likert scales from 0 to 10 to evaluate each use step ofthe medical device, closed-ended questions and open questions fr comments. It will be asked at the end of the clinical study at each caregiver.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Assistance Publique Hôpitaux de Paris, Hôpital Avicenne, Bobigny
  - Hôpital Louis Pradel, Bron
  - CHU Grenoble Alpes, Grenoble

REFERENCES:
- See also: Informations about CIC-IT — http://www.cic-it-grenoble.fr